CLINICAL TRIAL: NCT06932458
Title: A Phase II Single-arm Clinical Trial of Primary Retroperitoneal Lymph Node Dissection in Patients With Testicular Seminoma With Limited Retroperitoneal Metastases
Brief Title: A Clinical Trial of Primary Retroperitoneal Lymph Node Dissection in Patients With Testicular Seminoma With Limited Retroperitoneal Metastases
Acronym: RPLND-Seminoma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Western University, Canada (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 126353
Record Dates: First submitted 2025-04-09; First posted 2025-04-17 (Actual); Last update posted 2025-07-20 (Actual); Status verified 2025-07

CONDITIONS: Testicular Cancer
Keywords: Seminoma; Retroperitoneal lymph node dissection
MeSH Terms: conditions — Testicular Neoplasms; Seminoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CS IIA/IIB Seminoma (Other): Patients with relapsed CS I or de novo CS IIA/B with <3cm lymph node in the retroperitoneal lymph node.
  Interventions: Procedure: Retroperitoneal Lymph Node Dissection

INTERVENTIONS:
Procedure: Retroperitoneal Lymph Node Dissection — Open bilateral nerve-sparing RPLND.

SUMMARY:
Testicular cancer represents 1% of adult neoplasms and is the most common solid malignancy in young men. At diagnosis, approximately 90% of cases are germ cell tumours (GCT), categorised as either seminoma (55-60%) or non-seminoma types (40-45%).

For many years, the management of patients with CS IIA/B seminoma and retroperitoneal lymph node involvement ≤ 3 cm are eligible for treatment with either radiotherapy or chemotherapy Despite high cure rates for CS II seminoma (approximately 90%) with chemotherapy or radiotherapy, concerns persist regarding short and long-term treatment-related toxicities (such as increased risks of cardiovascular disease and secondary malignancies As such, an alternative strategy which has been explored in this study is the role of RPLND for the management of these patients

DETAILED DESCRIPTION:
Testicular cancer represents 1% of adult neoplasms and is the most common solid malignancy in young men. At diagnosis, approximately 90% of cases are germ cell tumours (GCT), categorised as either seminoma (55-60%) or non-seminoma types (40-45%). Approximately 20% of men with seminoma present with clinical stage (CS) II disease, characterized by enlarged retroperitoneal lymph nodes without distant metastasis.

For many decades for patients who recur following CS 1 seminoma or present with de novo CS IIA/B seminoma, either radiotherapy (30-36Gy) or chemotherapy (BEPx3, EPx4) has been the mainstay of treatment. Yet, both treatment paradigms carry significant short and long-term treatment-related toxicities. Radiotherapy, when compared to surveillance or surgery alone, has been shown to double the risk of cardiovascular disease and secondary malignancies (with an incidence of 2-3%). Additionally, patients who receive chemotherapy for GCTs can develop complications including irreversible neurotoxicity (10%), ototoxicity (5-12%), pulmonary toxicity, which may result in permanent restrictive lung disease (8%), metabolic syndrome (10-16%), and hypogonadism (4%). Additionally, patients are at an approximate 3-7-fold increase in cardiovascular mortality and a two-fold increase in secondary solid malignancies and leukaemia. Furthermore, both treatment modalities can harm fertility potential by approximately 20-30%.

However, in the past few years, a number of prospective single arm studies have been published evaluating the role of RPLND. RPLND is an appealing choice for patients with low-volume metastatic seminoma for several reasons: Firstly, seminoma exhibits a more indolent biological behaviour and a predictable lymphatic spread pattern compared to non-seminoma diseases, potentially allowing a greater chance of cure with surgery alone. Secondly, RPLND enables precise pathological staging which can avoid overtreatment in those with pathologically negative lymph nodes. It offers an opportunity to reduce the burden of chemotherapy by reserving this treatment only for the small proportion of men who will relapse following RPLND. Finally, RPLND offers an acceptably low risk of short or long-term complications when performed at experienced centres.

Therefore, our objective is to prospectively evaluate the short and long-term safety and efficacy of Primary Retroperitoneal Lymph Node Dissection (RPLND) for patients with testicular seminoma and limited retroperitoneal lymph node metastasis.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients (>18 years) with pure seminoma on radical orchiectomy specimen.
2. Initial CS I presentation with subsequent retroperitoneal relapse on surveillance, or de novo CS II at presentation.
3. Axial imaging of lymphadenopathy within 8 weeks of the date of RPLND

   1. No more than 2 enlarged retroperitoneal lymph nodes, each no more than 3cm in the primary landing zones.
   2. Suitable for proposed bilateral RPLND template
4. Serum tumour markers (alpha-fetoprotein (AFP), human chorionic gonadotropin (HCG), and lactate dehydrogenase (LDH)) must all be within normal limits within 2 weeks of planned RPLND

Exclusion Criteria:

1. Any condition deemed by the treating surgeon to pose an unacceptable risk for retroperitoneal lymph node dissection
2. Any non-seminoma component on the orchiectomy specimen.
3. AFP >20 at any time point, pre- or post-orchiectomy.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-07-17 (Estimated); Primary Completion 2028-06-01 (Estimated); Study Completion 2030-06-01 (Estimated)

PRIMARY OUTCOMES:
Recurrence Free Survival | 2 years
  2-year RFS (absence of radiological metastases on cross-sectional imaging and normal serum tumour markers).

SECONDARY OUTCOMES:
Complications | 90 days
  Complications post RPLND (Clavein-Dindo)
Length of Stay in hospital | 90 days
  Length of stay in hospital post RPLND
Treatment-Free Survival | 24 months
  Patients avoiding additional treatments for seminoma post RPLND (e.g. chemotherapy / radiotherapy)
Cancer-specific Survival | 24 months
  Percentage of people who have not died from testicular cancer during follow-up
Overall Survival | 2 years
  Patients alive during follow-up

CONTACTS AND LOCATIONS:
Locations (1):
- London Health Sciences Centre, London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Fung C, Dinh P Jr, Ardeshir-Rouhani-Fard S, Schaffer K, Fossa SD, Travis LB. Toxicities Associated with Cisplatin-Based Chemotherapy and Radiotherapy in Long-Term Testicular Cancer Survivors. Adv Urol. 2018 Feb 18;2018:8671832. doi: 10.1155/2018/8671832. eCollection 2018. PMID 29670654
- [Background] Fossa SD, Dahl AA, Thorsen L, Hellesnes R, Kiserud CE, Tandstad T, Brydoy M, Haugnes HS, Myklebust TA. Mortality and Second Cancer Incidence After Treatment for Testicular Cancer: Psychosocial Health and Lifestyle Are Modifiable Prognostic Factors. J Clin Oncol. 2022 Aug 10;40(23):2588-2599. doi: 10.1200/JCO.21.02105. Epub 2022 Apr 5. PMID 35380874
- [Background] Hamilton RJ, Canil C, Shrem NS, Kuhathaas K, Jiang MD, Chung P, North S, Czaykowski P, Hotte S, Winquist E, Kollmannsberger C, Aprikian A, Soulieres D, Tyldesley S, So AI, Power N, Rendon RA, O'Malley M, Wood L. Canadian Urological Association consensus guideline: Management of testicular germ cell cancer. Can Urol Assoc J. 2022 Jun;16(6):155-173. doi: 10.5489/cuaj.7945. No abstract available. PMID 35623007